CLINICAL TRIAL: NCT00628342
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Efficacy Study Comparing 4 Weeks of Treatment With Esomeprazole 20 mg qd and 40 mg qd to Placebo qd in Patients With Heartburn and Sleep Disturbances Associated With Gastroesophageal Reflux Disease (GERD)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Tore Lind, MD - Nexium Medical Science Director, AstraZeneca
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D961AC00001
Record Dates: First submitted 2008-02-26; First posted 2008-03-05 (Estimated); Last update posted 2009-03-12 (Estimated); Status verified 2009-03

CONDITIONS: Gastroesophageal Reflux Disease (GERD)
Keywords: Gastroesophageal Reflux Disease; GERD; Esomeprazole; Heartburn; Nexium
MeSH Terms: conditions — Gastroesophageal Reflux; Heartburn | interventions — Esomeprazole

ARMS (3):
- 1 (Experimental)
  Interventions: Drug: Esomeprazole
- 2 (Experimental)
  Interventions: Drug: Esomeprazole
- 3 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Esomeprazole — 20mg Oral tablet once daily
  Other Names: Nexium
  Arms: 1
Drug: Esomeprazole — 40mg Oral tablet once daily
  Other Names: Nexium
  Arms: 2
Drug: Placebo — Oral once daily
  Arms: 3

SUMMARY:
This study includes patients with sleep disturbances associated with gastroesophageal reflux disease (GERD) and has 3 treatment arms. Patients will receive only one of the following treatment arms: esomeprazole 20 mg once daily, esomeprazole 40 mg once daily, matching placebo once daily. The relief to the sleep disturbances will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* A history of heartburn or acid regurgitation for 3 months or longer or any history of erosive esophagitis.
* Nightime heartburn averaging at least 2 or 3 times per week and a history of sleep disturbances associated with GERD for 1 month or more.
* Nightime heartburn graded as moderate or severe on 3 of the last 7 days of the run-in period and sleep disturbances associated with GERD as documented in the run-in diary card on at least 3 of the last 7 days of the run-in period..

Exclusion Criteria:

* Any condition other than GERD that is either the primary cause of, or a significant contributor to the patients sleep disturbance.
* Shift workers who work between 12am (midnight) and 6am.
* Sleep medication, antihistamine, benzodiazepine, or anti-anxiety medication use that has not been stable for at least 3 months or is not expected to remain stable during the patients participation in the study.
* Other diseases / conditions as listed in the protocol.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2003-04; Primary Completion 2003-08 (Actual); Study Completion 2003-08 (Actual)

PRIMARY OUTCOMES:
Daily patient diary cards to demonstrate whether there is a difference in the relief of nighttime heartburn between esomeprazole 20 mg once daily (E20), and placebo once daily and between esomeprazole 40 mg once daily (E40) in patients with GERD. | Daily diary cards completed by the patients.

SECONDARY OUTCOMES:
To assess the impact of treatment with E20 versus placebo and E40 versus placebo on sleep disturbances associated with GERD as measured by:Change in global PSQI score; Complete resolution of sleep disturbances; Relief of sleep disturbances; Perc | Daily diary cards completed by the patients
To assess the impact of treatment with E20 versus placebo and E40 versus placebo on heartburn as measured by:Complete resolution of daytime heartburn; Complete resolution of nightime heartburn; Relief of daytime heartburn; Improvement in the fre | Daily diary cards completed by the patients.
To quantify the difference during 4 weeks of treatment between E20 and E40 in patients with GERD as measured by: - Relief of nightime heartburn - Relief of sleep disturbances associated with GERD | Daily diary cards completed by the patients.

CONTACTS AND LOCATIONS:
Overall Officials: Paula Fernstrom, Study Director — Nexium Global Product Director, AstraZeneca

REFERENCES:
- [Derived] Johnson DA, Le Moigne A, Hugo V, Nagy P. Rapid resolution of sleep disturbances related to frequent reflux: effect of esomeprazole 20 mg in two randomized, double-blind, controlled trials. Curr Med Res Opin. 2015 Feb;31(2):243-50. doi: 10.1185/03007995.2014.991818. Epub 2015 Jan 9. PMID 25478944